CLINICAL TRIAL: NCT02612129
Title: Arimoclomol Prospective Double-blind, Randomised, Placebo-controlled Study in Patients Diagnosed With Niemann-Pick Disease Type C
Brief Title: Arimoclomol Prospective Study in Participants Diagnosed With Niemann-Pick Disease Type C
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ZevraDenmark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-ORZY-NPC-002
Expanded Access: NCT04316637 (Available)
Record Dates: First submitted 2015-11-12; First posted 2015-11-23 (Estimated); Results first posted 2023-06-09 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Niemann-Pick Disease, Type C
Keywords: NPC1; Niemann-Pick Type C; Niemann-Pick; arimoclomol; lysosomal storage disorder; lysosomal storage disease; NPC2; NP-C
MeSH Terms: conditions — Niemann-Pick Disease, Type C; Lysosomal Storage Diseases | interventions — arimoclomol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arimoclomol Single PK Dose (Experimental): Participants less than 12 years received a single oral dose of arimoclomol capsule, based on participant's body weight, on Day 1.
  Interventions: Drug: arimoclomol
- Arimoclomol (12-month Double-blind Phase) (Experimental): Participants received arimoclomol capsules orally three times a day (TID) for 12 months. The dose was 31-124 mg arimoclomol base TID (equivalent to 50-200 mg arimoclomol citrate TID), based on participant's body weight.
  Interventions: Drug: arimoclomol
- Placebo (12-month Double-blind Phase) (Placebo Comparator): Participants received matching placebo capsules (with regard to weight, appearance, smell, flavor etc.) orally TID for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: arimoclomol
  Arms: Arimoclomol (12-month Double-blind Phase); Arimoclomol Single PK Dose
Drug: Placebo
  Arms: Placebo (12-month Double-blind Phase)

SUMMARY:
A prospective, randomized, double-blind, placebo controlled therapeutic study in participants with confirmed diagnosis of Niemann-Pick disease type C (NPC).

The purpose of this study is to assess the efficacy and safety of arimoclomol (compared to placebo) when it is administered as an add-on therapy to the participant's current prescribed best routine clinical care; participant's routine clinical care may, or may not, include miglustat.

The CT-ORZY-NPC-002 study has been expanded to include an open label paediatric sub-study including participants aged 6 to <24 months at study enrolment.

DETAILED DESCRIPTION:
A prospective, randomized, double-blind, placebo controlled therapeutic study in participants with confirmed diagnosis of Niemann-Pick disease type C (NPC).

Participants must either 1) have completed Visit 2 (end of study [EOS]) of the CT-ORZY-NPC-001 study or 2) meet the eligibility criteria of this study including a requirement of stable treatment with miglustat for 6 months (if on miglustat therapy) prior to enrolment into the study.

Aim:

The purpose of this study is to assess the efficacy and safety of arimoclomol (compared to placebo) when it is administered as an add-on therapy to the participant's current prescribed best routine clinical care; participant's routine clinical care may, or may not, include miglustat.

Randomization:

Participants will be randomized to receive placebo or arimoclomol (with an allocation ratio of 1:2).

Pharmacokinetic evaluation (age below 12):

To confirm the selected dose, participants less than 12 years of age will undergo an arimoclomol single-dose pharmacokinetic (PK) evaluation before randomization and the start of continuous (multiple dosing) treatment.

Early Escape Clause:

In participants whose disease progression is too severe and/or too fast, the "early escape clause" will allow the Investigator to apply the escape route which implies that the participant can be treated with arimoclomol (as per blinded phase study schedule) and be followed up according to the study schedule or until the analysis of data from the controlled, 12-month blinded phase study period does not support the efficacy and/or safety of arimoclomol.

Study duration:

The duration of the blinded phase study period will be 12-months.

Following this, all participants will be offered to continue into the extension phase of the study where every participant will receive arimoclomol and be followed up and attend site visits every 6 months until 60 months after randomization. The extension phase runs until arimoclomol has received Regulatory Approval or until the analysis of data from the controlled, blinded phase 12-month study period does not support the efficacy and/or safety of arimoclomol.

The CT-ORZY-NPC-002 protocol has been updated to include a paediatric sub-study including new and naïve participants aged 6 to <24 months at study enrolment.

Aim:

The purpose of the paediatric sub-study, is to assess the safety and tolerability of 36 months of open-label arimoclomol when administered as an add-on therapy to the participant's current prescribed best routine clinical care; participant's routine clinical care may, or may not, include miglustat.

The Paediatric sub-study will run at the open sites participating in the main study. A total of 3-5 participants are planned to be enrolled. All participants will be treated with arimoclomol.

Main Inclusion Criteria:

* Diagnosis of NPC1 or NPC2;
* NPC diagnosis confirmed by:

  * Genetically confirmed (deoxyribonucleic acid [DNA] sequence analysis) by mutations in both alleles of NPC1 or NPC2, OR
  * Mutation in only one allele of NPC1 or NPC2 plus either positive filipin staining or elevated cholestane triol/oxysterols (>2 x upper limit of normal).
* Males and females aged 6 to <24 months, with a cap of maximum 3 participants above 18 months
* Treated or not treated with miglustat;

  * If a participant is on prescribed treatment with miglustat, the dose must have been stable for at least 1 month prior to inclusion in the paediatric sub-study
  * If a participant has been discontinued from prescribed treatment with miglustat, they must have been discontinued for at least 1 month prior to inclusion in the paediatric sub-study
* The Legal Authorised Representative (LAR) has read and signed the Informed Consent Form (ICF) prior to any study-related procedures
* The LAR agrees for the participant to participate in all aspects of the trial design

Main Exclusion Criteria:

* Recipient of a liver transplant or a planned liver transplant
* The Aspartate Transaminase (AST) and/or Alanine Transaminase (ALT) >3 x Upper Limit of Normal (ULN) for age and gender
* Renal insufficiency with serum creatinine level >1.5 x ULN
* Participants with known causes of active liver disease or prolonged icterus or malformation of organs other than NPC
* Participant was born before 37 weeks of gestation
* Participant weight <5 kg at study enrollment
* Participant is diagnosed with severe intra-uterine growth restriction
* Participant has severe neurological symptoms
* Participant has received or plans to receive a bone marrow transplant

Arms and Intervention:

1 arm open label treatment with arimoclomol capsules 100 mg (dispersed in water) for oral administration (3 times daily). Doses: The dose in mL is based on the participant's weight in kg.

Randomization: Open Label

Pharmacokinetic: To confirm the selected dose, participants will undergo an arimoclomol single-dose pharmacokinetic (PK) evaluation before the start of continuous treatment.

Visit schedule time frame: Screening (V1); enrollment Week 1 (V2 baseline), Weeks 2 (V3), continuing visits at months 1 (V4), 3 (V5), 6 (V6), 9 (V7), 12 (V8), 15 (V8a), 18 (V9), 24 (V10), 30 (V11) and 36 (V12).

Primary objective: Safety and tolerability

Main Endpoint measures:

Safety data: Adverse events (AEs); Vital signs; Hematology; Clinical chemistry

Clinical status data: Clinical signs and symptoms captured through physical examination; Change from baseline in patient weight and height; Change in Bayley III score: Developmental delay scoring

Imaging data: Changes from baseline in the size of the liver and spleen assessed by ultrasound

ELIGIBILITY:
Inclusion Criteria:

EITHER NP-C participants who have entered the CT-ORZY-NPC-001 study and who have completed Visit 2 (EOS) of the CT-ORZY-NPC-001 study.

OR

NPC participants who did not enter or complete the CT-ORZY-NPC-001 study but are fulfilling all of criteria listed below:

◦Diagnosis of NPC1 or NPC2;

NPC diagnosis confirmed by:

* Genetically confirmed (deoxyribonucleic acid [DNA] sequence analysis) by mutations in both alleles of NPC1 or NPC2, OR
* Mutation in only one allele of NPC1 or NPC2 plus either positive filipin staining or elevated cholestane triol/oxysterols (>2 x upper limit of normal).

  * Males and females aged from 2 years to 18 years and 11 months;
  * Treated or not treated with miglustat;
  * If a participant is under prescribed treatment with miglustat, it has to be under stable dose of the medication for at least 6 continuous months prior to inclusion in the CT-ORZY-NPC-002 study;

    o If a participant has been discontinued from prescribed treatment with miglustat, they must have been discontinued for at least 3 continuous months prior to inclusion in the CT-ORZY-NPC-002 study;
  * Body mass index (BMI) Z score ≥ -2 SD (standard deviation) for age, according to the World Health Organisation (WHO) standards;
  * Presenting at least one neurological symptom of the disease (for example, but not limited to, hearing loss, vertical supranuclear gaze palsy, ataxia, dementia, dystonia, seizures, dysarthria, or dysphagia);
  * Ability to walk either independently or with assistance.

    * Written informed consent (and assent if appropriate to local laws and regulations) prior to any study-related procedures;
    * Willing to participate in all aspects of trial design including blood sampling (PK, blood biomarkers and safety labs), skin biopsies and imaging (ultrasonography of the liver and spleen);
    * Ability to travel to the corresponding clinical trial site at the scheduled visit times for evaluation and follow-up;
    * All sexually active female participants of child-bearing potential (post-menarchal) must use highly effective contraception during the study and until 1 week after the last dose of IMP.

Highly effective birth control methods include: Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable); intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; and vasectomised partner.

All sexually active male participants with female partners of child-bearing potential (post-menarchal) must use a condom with or without spermicide in addition to the birth control used by their partners during the study and until 3 months after the last dose of IMP.

Sexual abstinence is considered a highly effective birth control method only if it is defined as refraining from heterosexual intercourse during the study and for 1 week after the last dose of IMP (for female participants of child-bearing potential) and for 3 months after the last dose of IMP (for male participants with female partners of child-bearing potential). The reliability of sexual abstinence needs to be evaluated by the Investigator in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant.

•Ability to comply with the protocol-specified procedures/evaluations and scheduled visits.

Exclusion Criteria:

* Recipient of a liver transplant or planned liver transplantation;
* Severe liver insufficiency (defined as hepatic laboratory parameters, AST and/or ALT greater than three-times the upper limit of normal for age and gender (central laboratory assessment);
* Renal insufficiency, with serum creatinine level greater than 1.5 times the upper limit of normal (central laboratory assessment);
* Known or suspected allergy or intolerance to the IMP (arimoclomol or constituents);
* In the opinion of the Investigator, the participant's clinical condition does not allow for the required blood collection and/or skin biopsies as per the protocol-specified procedures;
* Treatment with any investigational drug during the study or in the 4 weeks prior to entering the study.

This includes treatment with any investigational drug during the study in an attempt to treat NP-C;

* Pregnancy or breastfeeding;
* Current participation in another trial is not permitted unless it is a non-interventional study and the sole purpose of the trial is for long-term follow up/survival data (registry);
* For participants who have not completed the CT-ORZY-NPC-001 study, fulfilling any of the criteria listed below:

  * Participants with uncontrolled severe epileptic seizures period (at least 3 consecutive severe epileptic seizures that required medication) within 2 months prior to the written consent. This includes participants with ongoing seizures that are not stable in frequency or type or duration over a 2 month period prior to enrolment, requiring change in dose of antiepileptic medication (other than adjustment for weight) over a 2 month period prior to enrolment, or requiring 3 or more antiepileptic medications to control seizures;
  * Neurologically asymptomatic participants;
  * Severe manifestations of NP-C disease that would interfere with the participant's ability to comply with the requirements of this protocol;
  * Treatment with any IMP within 4 weeks prior to the study enrolment.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Eugen Mengel, Principal Investigator — SphinCS GmbH, Hochheim, Germany
Locations (14):
- United States (2):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Mayo Clinic Children's Center, Rochester, Minnesota
- University Hospital Copenhagen (Rigshospitalet), Copenhagen, Denmark
- France (2):
  - CHU de Montpellier, Montpellier
  - Hôpital Trousseau, Paris
- Germany (2):
  - Villa Metabolica, Universitätsmedizin Mainz, Mainz
  - Dr. von Haunersches Kinderspital der Universität München, Munich
- Italy (2):
  - Ospedale Pediatrico Bambino Gesù, Rome
  - Azienda Ospedaliero-Universitaria "Santa Maria della Misericordia" di Udin, Udine
- The Children´s Memorial Istitute Warsaw, Warsaw, Poland
- Hospital Vall D'Hebron, Barcelona, Spain
- INSELSPITAL University Hospital Bern, Bern, Switzerland
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham
  - Great Ormond Street Hospital, London

REFERENCES:
- [Background] Patterson MC, Lloyd-Price L, Guldberg C, Doll H, Burbridge C, Chladek M, iDali C, Mengel E, Symonds T. Validation of the 5-domain Niemann-Pick type C Clinical Severity Scale. Orphanet J Rare Dis. 2021 Feb 12;16(1):79. doi: 10.1186/s13023-021-01719-2. PMID 33579322
- [Result] Mengel E, Patterson MC, Da Riol RM, Del Toro M, Deodato F, Gautschi M, Grunewald S, Gronborg S, Harmatz P, Heron B, Maier EM, Roubertie A, Santra S, Tylki-Szymanska A, Day S, Andreasen AK, Geist MA, Havnsoe Torp Petersen N, Ingemann L, Hansen T, Blaettler T, Kirkegaard T, I Dali C. Efficacy and safety of arimoclomol in Niemann-Pick disease type C: Results from a double-blind, randomised, placebo-controlled, multinational phase 2/3 trial of a novel treatment. J Inherit Metab Dis. 2021 Nov;44(6):1463-1480. doi: 10.1002/jimd.12428. Epub 2021 Sep 7. PMID 34418116

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 14 sites in Denmark, France, Germany, Italy, Poland, Spain, Switzerland, United Kingdom, and United States.
Pre-assignment Details: To confirm the selected dose of arimoclomol for participants less than 12 years of age, the 28 participants below 12 years old received a single arimoclomol dose for PK evaluation before randomization and the start of continuous treatment. A total of 50 participants were randomized in the blinded phase (continuous dose phase) and the study is ongoing in an open-label period.
Groups:
- Arimoclomol (12-month Double-blind Phase): Participants received arimoclomol capsules, orally based on participant's body weight, three times a day (TID) for 12 months.
- Placebo (12-month Double-blind Phase): Participants received matching placebo to arimoclomol capsules, orally based on participant's body weight, TID for 12 months.
Period: Single Dose Treatment Period
Arm/Group | Arimoclomol Single PK Dose | Arimoclomol (12-month Double-blind Phase) | Placebo (12-month Double-blind Phase)
Started | 28 | 0 | 0
Completed (One participant who was a screening failure received single-dose arimoclomol for PK evaluation.) | 27 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Screening Failure | 1 | 0 | 0
Period: Continuous Treatment Period
Arm/Group | Arimoclomol Single PK Dose | Arimoclomol (12-month Double-blind Phase) | Placebo (12-month Double-blind Phase)
Started | 0 | 34 | 16
Completed | 0 | 27 | 15
Not Completed | 0 | 7 | 1
Not completed — Early Escape | 0 | 2 | 0
Not completed — Participant's Parents/legal guardian have Withdrawn Informed Consent | 0 | 1 | 0
Not completed — Safety Reasons | 0 | 3 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Participant Meets Criteria for IMP Administration to be Stopped and Subsequent Withdrawal | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included those participants who were randomized and who had received at least one dose of randomized treatment medication.
Groups:
- Arimoclomol (12-month Double-blind Phase): Participants received arimoclomol capsules, orally based on participant's body weight, TID for 12 months.
- Total: Total of all reporting groups
Arm/Group | Arimoclomol (12-month Double-blind Phase) | Placebo (12-month Double-blind Phase) | Total
Number analyzed (Participants) | 34 | 16 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.5 (5.4) | 10.2 (4.1) | 11.1 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 26
  Male | 17 | 7 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 32 | 16 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 32 | 13 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Age at Diagnosis of First Neurological Symptom [Mean (Standard Deviation); unit: years] | 5.05 (3.43) | 5.22 (3.87) | 5.10 (3.54)
5-domain Niemann-Pick Disease Type C Clinical Severity Scale (NPCCSS) Score [Mean (Standard Deviation); unit: score on a scale] — The 5-domain NPC Clinical Severity Scale (NPCCSS) focuses on domains identified by participants, caregivers, and NPC experts as the most clinically relevant when assessing disease progression in NPC: Ambulation, fine motor skills, swallow, cognition, and speech. The scale is derived from the original 17-domain NPCCSS. Each domain is rated on a scale of 0-5 based on clinical assessments, observations, and interviews with participants/caregiver. The total score is a sum of the score of each of the 5 domains and ranges from 0-25, with a higher score indicating more severe clinical impairment.
  score on a scale | 12.1 (6.9) | 9.4 (6.4) | 11.2 (6.8)
17-domain NPCCSS Except Hearing Domains [Mean (Standard Deviation); unit: score on a scale] — The NPC Clinical Severity Scale (NPCCSS) is a disease-specific, clinician-reported outcome measure developed to characterize and quantify NPC disease progression. The 17-domain NPCCSS includes clinical signs and symptoms in nine major and eight minor domains, which are rated on scales of 0-5 (for the major domains) or 0-2 (for the minor domains). The total score is the sum of the score of each of the 17 domains and ranges from 0 to 61, with a high score indicating a more severe clinical impairment.
  score on a scale | 21.2 (11.5) | 17.2 (11.3) | 19.9 (11.4)
Participants Currently Treated With Miglustat [Count of Participants; unit: Participants]
  Yes | 26 | 13 | 39
  No | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Niemann-Pick Disease Type C (NPC) Disease Severity Assessed Based on the 5-domain NPCCSS Total Scores
Description: NPC disease severity was assessed based on the 5-domain NPC Clinical Severity Scale (NPCCSS). The 5-domain NPCCSS focuses on domains identified by participants, caregivers, and NPC experts as the most clinically relevant when assessing disease progression in NPC: Ambulation, fine motor skills, swallow, cognition, and speech. The scale is derived from the original 17-domain NPCCSS. Each domain is rated on a scale of 0-5 based on clinical assessments, observations, and interviews with participants/caregiver. The total score is a sum of the score of each of the 5 domains and ranges from 0-25, with a higher score indicating more severe clinical impairment.
Time Frame: Baseline to Month 12
Population: Full Analysis Set (FAS) included those participants who were randomized and who had received at least one dose of randomized treatment medication. Overall Number analyzed is the number of participants evaluated at a specified timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arimoclomol (12-month Double-blind Phase) | Placebo (12-month Double-blind Phase)
Number analyzed (Participants) | 27 | 15
score on a scale | 0.76 [-0.05 to 1.56] | 2.15 [1.05 to 3.25]
Statistical Analysis 1: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); A general linear mixed model (GLMM) for repeated measurements was used for the analysis of NPC disease severity assessed based on the 5-domain NPCCSS scores at Month 12. The general linear mixed model analysis for repeated measures was fitted with treatment, miglustat level and visit as fixed effects including treatment-by-visit interaction and baseline score as a covariate; Test type: Superiority; p = 0.0456, GLMM for Repeated Measures; Least Square (LS) Mean Difference = -1.40, 95% CI 2-sided [-2.76 to -0.03]

2. Secondary Outcome: Percentage of Responders in Clinical Global Impression Scale of Improvement (CGI-I) - Defined as Percentage of Participants Where the CGI-I Score Remains Stable or Shows Improvement (This Outcome Measure Was Considered Co-primary by the FDA)
Description: The CGI-I is a 7-point scale that rates total improvement of participant's condition. The clinician rates the participants from 1=Very much improved, 2=Much improved, 3=Minimally improved, 4=No change, 5=Minimally worse, 6=Much worse, or 7=Very much worse. Scores thus range from 1-7 with lower scores indicating greater improvement. Responders were the participants with a score of 1 or 2 at Month 12.
Time Frame: Month 12
Population: FAS included those participants who were randomized and who had received at least one dose of randomized treatment medication.
Measure: Number; unit: percentage of responders
Arm/Group | Arimoclomol (12-month Double-blind Phase) | Placebo (12-month Double-blind Phase)
Number analyzed (Participants) | 34 | 16
percentage of responders | 58.8 | 56.3
Statistical Analysis 1: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Test type: Superiority; p = 1.0000, Chi-squared Test

3. Secondary Outcome: Percentage of Responders in 5-domain NPCCSS - Defined as Participants Where the 5-domain NPCCSS Score Remains Stable or Improves as Compared to Baseline
Description: NPC disease severity was assessed based on the 5-domain NPC Clinical Severity Scale (NPCCSS). The 5-domain NPCCSS focuses on domains identified by participants, caregivers, and NPC experts as the most clinically relevant when assessing disease progression in NPC: Ambulation, fine motor skills, swallow, cognition, and speech. The scale is derived from the original 17-domain NPCCSS. Each domain is rated on a scale of 0-5 based on clinical assessments, observations, and interviews with participants/caregiver. The total score is a sum of the score of each of the 5 domains and ranges from 0-25, with a higher score indicating more severe clinical impairment. Stable was defined as a participant's total score for the 5 domains being the same at month 12 as at baseline. Improvement was defined as a participant's total score at month 12 being lower than at baseline.
Time Frame: Baseline to Month 12
Population: as for outcome 2
Measure: Number; unit: percentage of responders
Arm/Group | Arimoclomol (12-month Double-blind Phase) | Placebo (12-month Double-blind Phase)
Number analyzed (Participants) | 34 | 16
percentage of responders | 50.0 | 37.5
Statistical Analysis 1: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Test type: Superiority; p = 0.5456, Chi-squared Test

4. Secondary Outcome: Time to Worsening
Description: Time to worsening was defined as the time until the participant reached the predefined minimal clinically important difference (MCID) of 2 points compared to baseline on the 5-domain NPC Clinical Severity Scale (NPCCSS). The 5-domain NPCCSS focuses on domains identified by participants, caregivers, and NPC experts as the most clinically relevant when assessing disease progression in NPC: Ambulation, fine motor skills, swallow, cognition, and speech. The scale is derived from the original 17-domain NPCCSS. Each domain is rated on a scale of 0-5 based on clinical assessments, observations, and interviews with participants/caregiver. The total score is a sum of the score of each of the 5 domains and ranges from 0-25, with a higher score indicating more severe clinical impairment. The values reported per group are the 25th percentile Kaplan-Meier estimates and 95% confidence interval.
Time Frame: Baseline to Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Arimoclomol (12-month Double-blind Phase) | Placebo (12-month Double-blind Phase)
Number analyzed (Participants) | 34 | 16
months | 5.2 [2.9 to 12.0] | 5.5 [1.0 to 6.5]
Statistical Analysis 1: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Log-rank test had been stratified by miglustat use; Test type: Superiority; p = 0.8021, Log-Rank Test

5. Secondary Outcome: Percentage of Participants With Worsening
Description: Worsening was defined as participants that have reached the predefined MCID of 2 points on their 5-domain NPC Clinical Severity Scale (NPCCSS). The 5-domain NPCCSS focuses on domains identified by participants, caregivers, and NPC experts as the most clinically relevant when assessing disease progression in NPC: Ambulation, fine motor skills, swallow, cognition, and speech. The scale is derived from the original 17-domain NPCCSS. Each domain is rated on a scale of 0-5 based on clinical assessments, observations, and interviews with participants/caregiver. The total score is a sum of the score of each of the 5 domains and ranges from 0-25, with a higher score indicating more severe clinical impairment.
Time Frame: Months 6 and 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Arimoclomol (12-month Double-blind Phase) | Placebo (12-month Double-blind Phase)
Number analyzed (Participants) | 34 | 16
percentage of participants
  Worsening at Month 6 | 35.3 | 50.0
  Worsening at Month 12 | 44.1 | 43.8
Statistical Analysis 1: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Percentage of participants worsening at Month 6; Test type: Superiority; p = 0.3662, Fisher's Exact Test
Statistical Analysis 2: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Percentage of participants worsening at Month 12; Test type: Superiority; p = 1.0000, Fisher's Exact Test

6. Secondary Outcome: Change From Baseline in 17-domain NPCCSS Apart From Hearing Domains (i.e. Hearing and Auditory Brainstem Response)
Description: The NPC Clinical Severity Scale (NPCCSS) is a disease-specific, clinician-reported outcome measure developed to characterize and quantify NPC disease progression. The 17-domain NPCCSS includes clinical signs and symptoms in nine major and eight minor domains, which are rated on scales of 0-5 (for the major domains) or 0-2 (for the minor domains). The total score is the sum of the score of each of the 17 domains and ranges from 0 to 61, with a high score indicating a more severe clinical impairment.
Time Frame: Baseline to 6 and 12 months
Population: FAS included those participants who were randomized and who had received at least one dose of randomized treatment medication. Here, "Number analyzed" signifies number of participants evaluated at specified timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arimoclomol (12-month Double-blind Phase) | Placebo (12-month Double-blind Phase)
Number analyzed (Participants) | 34 | 16
score on a scale
  Change at Month 6 | 0.53 [-0.85 to 1.90] | 2.22 [0.33 to 4.10]
  Change at Month 12 | 1.20 [-0.40 to 2.79] | 2.81 [0.75 to 4.87]
Statistical Analysis 1: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Change From Baseline in 17-Domain NPCCSS Apart from Hearing Domains (i.e. Hearing and Auditory Brainstem Response) at Month 6 was analyzed using the Analysis of covariance (ANCOVA) model. ANCOVA model was fitted with treatment, baseline full-scale NPCCSS apart from hearing domains score, and use of miglustat as covariates; Test type: Superiority; p = 0.1546, ANCOVA; LS Mean Difference = -1.69, 95% CI 2-sided [-4.04 to 0.66]
Statistical Analysis 2: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Change From Baseline in 17-Domain NPCCSS Apart from Hearing Domains (i.e. Hearing and Auditory Brainstem Response) at Month 12 was analyzed using the ANCOVA model. ANCOVA model is fitted with treatment, baseline full-scale NPCCSS apart from hearing domains score, and use of miglustat as covariates; Test type: Superiority; p = 0.2199, ANCOVA; LS Mean Difference = -1.61, 95% CI 2-sided [-4.24 to 1.01]

7. Secondary Outcome: Change From Baseline in 5-domain NPCCSS Score
Description: The 5-domain NPC Clinical Severity Scale (NPCCSS) focuses on domains identified by participants, caregivers, and NPC experts as the most clinically relevant when assessing disease progression in NPC: Ambulation, fine motor skills, swallow, cognition, and speech. The scale is derived from the original 17-domain NPCCSS. Each domain is rated on a scale of 0-5 based on clinical assessments, observations, and interviews with participants/caregiver. The total score is a sum of the score of each of the 5 domains and ranges from 0-25, with a higher score indicating more severe clinical impairment.
Time Frame: Baseline to 6 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arimoclomol (12-month Double-blind Phase) | Placebo (12-month Double-blind Phase)
Number analyzed (Participants) | 34 | 16
score on a scale | 0.48 [-0.05 to 1.02] | 1.60 [0.86 to 2.34]
Statistical Analysis 1: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); An ANCOVA model was fitted with treatment, baseline 5-domain NPCCSS score, and use of miglustat as covariates; Test type: Superiority; p = 0.0188, ANCOVA; Least Square (LS) Mean Difference = -1.11, 95% CI 2-sided [-2.03 to -0.19]

8. Secondary Outcome: Changes From Baseline in Each Individual Domain of the NPCCSS
Description: The NPC Clinical Severity Scale (NPCCSS) is a disease-specific, clinician-reported outcome measure developed to characterize and quantify disease progression. The 17-domain NPCCSS includes clinical signs and symptoms in nine major (ambulation, cognition, eye movement, fine motor, hearing, memory, seizures, speech, swallowing,) and eight minor (auditory brainstem response, behavior, gelastic cataplexy, hyperreflexia, incontinence, narcolepsy, psychiatric, respiratory problems) domains, which are rated on scales of 0-5 (for the major domains) or 0-2 (for the minor domains). A higher score indicates a more severe clinical impairment.
Time Frame: Baseline to 6 and 12 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arimoclomol (12-month Double-blind Phase) | Placebo (12-month Double-blind Phase)
Number analyzed (Participants) | 34 | 16
score on a scale
  Ambulation: Baseline | 2.5 (1.6) | 2.2 (1.6)
  Ambulation: Change at Month 6: number analyzed (Participants) | 29 | 15
  Ambulation: Change at Month 6 | 0.1 (0.4) | 0.3 (1.0)
  Ambulation: Change at Month 12: number analyzed (Participants) | 27 | 15
  Ambulation: Change at Month 12 | 0.3 (0.5) | 0.3 (0.9)
  Speech: Baseline | 2.2 (1.6) | 1.6 (1.2)
  Speech: Change at Month 6: number analyzed (Participants) | 29 | 15
  Speech: Change at Month 6 | 0.1 (0.5) | 0.1 (0.3)
  Speech: Change at Month 12: number analyzed (Participants) | 27 | 15
  Speech: Change at Month 12 | -0.2 (1.0) | 0.3 (0.8)
  Swallow: Baseline | 1.9 (1.7) | 1.3 (1.7)
  Swallow: Change at Month 6: number analyzed (Participants) | 29 | 15
  Swallow: Change at Month 6 | 0.1 (1.1) | 0.4 (1.0)
  Swallow: Change at Month 12: number analyzed (Participants) | 27 | 15
  Swallow: Change at Month 12 | 0.1 (1.1) | 0.6 (1.0)
  Fine Motor Skills: Baseline | 2.8 (1.8) | 1.9 (1.8)
  Fine Motor Skills: Change at Month 6: number analyzed (Participants) | 29 | 15
  Fine Motor Skills: Change at Month 6 | 0.1 (0.7) | 0.5 (1.1)
  Fine Motor Skills: Change at Month 12: number analyzed (Participants) | 27 | 15
  Fine Motor Skills: Change at Month 12 | 0.2 (0.8) | 0.6 (1.3)
  Cognition: Baseline | 2.8 (1.3) | 2.5 (1.5)
  Cognition: Change at Month 6: number analyzed (Participants) | 29 | 15
  Cognition: Change at Month 6 | 0.2 (0.5) | 0.3 (0.8)
  Cognition: Change at Month 12: number analyzed (Participants) | 27 | 15
  Cognition: Change at Month 12 | 0.3 (0.6) | 0.1 (0.6)
  Eye Movement: Baseline | 2.2 (1.2) | 2.1 (1.1)
  Eye Movement: Change at Month 6: number analyzed (Participants) | 29 | 15
  Eye Movement: Change at Month 6 | 0.0 (0.6) | -0.1 (0.7)
  Eye Movement: Change at Month 12: number analyzed (Participants) | 27 | 15
  Eye Movement: Change at Month 12 | 0.2 (0.9) | -0.1 (0.6)
  Memory: Baseline: number analyzed (Participants) | 33 | 16
  Memory: Baseline | 1.9 (1.4) | 1.3 (1.5)
  Memory: Change at Month 6: number analyzed (Participants) | 28 | 15
  Memory: Change at Month 6 | 0.1 (0.5) | 0.2 (1.1)
  Memory: Change at Month 12: number analyzed (Participants) | 25 | 15
  Memory: Change at Month 12 | 0.1 (0.5) | 0.3 (0.8)
  Seizures: Baseline | 1.9 (1.9) | 1.3 (1.8)
  Seizures: Change at Month 6: number analyzed (Participants) | 29 | 15
  Seizures: Change at Month 6 | -0.1 (0.8) | 0.0 (1.5)
  Seizures: Change at Month 12: number analyzed (Participants) | 27 | 15
  Seizures: Change at Month 12 | 0.3 (0.8) | -0.1 (1.7)
  Hearing: Baseline: number analyzed (Participants) | 18 | 10
  Hearing: Baseline | 0.4 (1.0) | 0.0 (0.0)
  Hearing: Change at Month 6: number analyzed (Participants) | 13 | 7
  Hearing: Change at Month 6 | -0.2 (0.8) | 0.0 (0.0)
  Hearing: Change at Month 12: number analyzed (Participants) | 10 | 6
  Hearing: Change at Month 12 | 0.0 (0.0) | 0.3 (0.8)
  Auditory Brainstem Response: Baseline: number analyzed (Participants) | 10 | 7
  Auditory Brainstem Response: Baseline | 0.2 (0.4) | 0.1 (0.4)
  Auditory Brainstem Response: Change at Month 6: number analyzed (Participants) | 5 | 5
  Auditory Brainstem Response: Change at Month 6 | 0.0 (0.0) | 0.2 (0.4)
  Auditory Brainstem Response: Change at Month 12: number analyzed (Participants) | 5 | 5
  Auditory Brainstem Response: Change at Month 12 | 0.0 (0.0) | 0.0 (0.0)
  Behavior: Baseline | 0.4 (0.6) | 0.4 (0.6)
  Behavior: Change at Month 6: number analyzed (Participants) | 29 | 15
  Behavior: Change at Month 6 | 0.0 (0.5) | -0.1 (0.5)
  Behavior: Change at Month 12: number analyzed (Participants) | 27 | 15
  Behavior: Change at Month 12 | 0.1 (0.6) | -0.2 (0.4)
  Gelastic Cataplexy: Baseline | 0.8 (0.9) | 0.4 (0.8)
  Gelastic Cataplexy: Change at Month 6: number analyzed (Participants) | 29 | 15
  Gelastic Cataplexy: Change at Month 6 | 0.1 (0.5) | 0.3 (0.6)
  Gelastic Cataplexy: Change at Month 12: number analyzed (Participants) | 27 | 15
  Gelastic Cataplexy: Change at Month 12 | 0.2 (0.6) | 0.3 (0.6)
  Hyperreflexia: Baseline | 1.0 (0.7) | 1.1 (0.9)
  Hyperreflexia: Change at Month 6: number analyzed (Participants) | 29 | 15
  Hyperreflexia: Change at Month 6 | -0.0 (0.5) | 0.2 (0.6)
  Hyperreflexia: Change at Month 12: number analyzed (Participants) | 27 | 15
  Hyperreflexia: Change at Month 12 | 0.1 (0.7) | 0.1 (0.5)
  Incontinence: Baseline | 1.0 (0.8) | 0.8 (0.9)
  Incontinence: Change at Month 6: number analyzed (Participants) | 29 | 15
  Incontinence: Change at Month 6 | -0.1 (0.4) | 0.1 (0.5)
  Incontinence: Change at Month 12: number analyzed (Participants) | 27 | 15
  Incontinence: Change at Month 12 | -0.0 (0.4) | 0.1 (0.9)
  Narcolepsy (NARCO): Baseline | 0.1 (0.4) | 0.3 (0.7)
  Narcolepsy (NARCO): Change at Month 6: number analyzed (Participants) | 29 | 15
  Narcolepsy (NARCO): Change at Month 6 | 0.0 (0.4) | -0.1 (0.3)
  Narcolepsy (NARCO): Change at Month 12: number analyzed (Participants) | 27 | 15
  Narcolepsy (NARCO): Change at Month 12 | -0.1 (0.4) | -0.1 (0.3)
  Psychiatric: Baseline | 0.1 (0.4) | 0.1 (0.5)
  Psychiatric: Change at Month 6: number analyzed (Participants) | 29 | 15
  Psychiatric: Change at Month 6 | -0.0 (0.3) | 0.1 (0.6)
  Psychiatric: Change at Month 12: number analyzed (Participants) | 27 | 15
  Psychiatric: Change at Month 12 | 0.0 (0.3) | 0.0 (0.4)
  Respiratory: Baseline | 0.1 (0.3) | 0.0 (0.0)
  Respiratory: Change at Month 6: number analyzed (Participants) | 29 | 15
  Respiratory: Change at Month 6 | 0.0 (0.5) | 0.1 (0.3)
  Respiratory: Change at Month 12: number analyzed (Participants) | 27 | 15
  Respiratory: Change at Month 12 | 0.1 (0.5) | 0.2 (0.4)

9. Secondary Outcome: Change From Baseline in the NPC Clinical Database (NPC-CDB) Score (Modified "Stampfer Score")
Description: The NPC Clinical Database (NPC-cdb) score aims to reflect the current clinical status of the participant. The NPC-cdb score represents both historical symptoms and a current status. The test consists of ten areas: visceral signs, development, motor function, ocular-motor abnormalities, seizures/cataplexy/narcolepsy, cognitive abilities and memory, behavioral and psychiatric abnormalities, speech, hearing, and abilities in daily life. The current status score is a severity-weighted sum of 72 symptoms considered as disease-relevant at the time of assessment. Each symptom contributes with a score between 1 and 5, the maximum score is 125. An increase in score reflects a reduction in the participant's abilities.
Time Frame: Baseline to 6 and 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arimoclomol (12-month Double-blind Phase) | Placebo (12-month Double-blind Phase)
Number analyzed (Participants) | 34 | 16
score on a scale
  Change at Month 6 | -0.38 [-3.30 to 2.54] | 4.71 [0.49 to 8.93]
  Change at Month 12 | 1.85 [-2.16 to 5.86] | 4.88 [-0.63 to 10.39]
Statistical Analysis 1: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Change from baseline in the NPC-CDB score (modified "Stampfer Score") at Month 6 was analyzed using the ANCOVA model. ANCOVA model was fitted with treatment, baseline NPC-CDB total score and use of miglustat as covariates; Test type: Superiority; p = 0.0536, ANCOVA; LS Mean Difference = -5.09, 95% CI 2-sided [-10.26 to 0.08]
Statistical Analysis 2: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Change from baseline in the NPC-CDB score (modified "Stampfer Score") at Month 12 was analyzed using the ANCOVA model. ANCOVA model was fitted with treatment, baseline NPC-CDB total score and use of miglustat as covariates; Test type: Superiority; p = 0.3785, ANCOVA; LS Mean Difference = -3.03, 95% CI 2-sided [-9.90 to 3.85]

10. Secondary Outcome: Percentage of Participants With Change From Baseline in Quality of Life (EQ-5D-Y)
Description: The EQ-5D-Y descriptive system includes 5 descriptive items: Mobility, self-care, doing usual activities, having pain or discomfort, and feeling anxiety or depressed. Each dimension has 3 levels: No problems, some problems, and a lot of problems. The change in the 5 individual items of the EQ-5D-Y per participant was explored by using the pareto principle at 6 and 12 months to show the number (%) of participants who felt:
  * Better (better on at least one dimension and no worse in any other dimension),
  * Worse (worse in at least one dimension, and no better in any other dimension)
Time Frame: Baseline to 6 and 12 months
Population: FAS included those participants who were randomized and who had received at least one dose of randomized treatment medication. Here, "Overall Number of Participants Analyzed" is the number of participants with data for the outcome measure and "Number analyzed" signifies number of participants evaluated at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Arimoclomol (12-month Double-blind Phase) | Placebo (12-month Double-blind Phase)
Number analyzed (Participants) | 30 | 15
percentage of participants
  Better: Change at Month 6 | 16.7 | 26.7
  Worse: Change at Month 6 | 40.0 | 46.7
  Better: Change at Month 12: number analyzed (Participants) | 27 | 15
  Better: Change at Month 12 | 25.9 | 40.0
  Worse: Change at Month 12: number analyzed (Participants) | 27 | 15
  Worse: Change at Month 12 | 44.4 | 20.0
Statistical Analysis 1: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Percentage of participants with change from baseline at Month 6 in Quality of Life (EQ-5D-Y) being 'Better'; Test type: Superiority; p = 0.6951, Chi-squared Test
Statistical Analysis 2: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Percentage of participants with change from baseline at Month 6 in Quality of Life (EQ-5D-Y) being 'Worse'; Test type: Superiority; p = 0.7542, Chi-squared Test
Statistical Analysis 3: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Percentage of participants with change from baseline at Month 12 in Quality of Life (EQ-5D-Y) being 'Better'; Test type: Superiority; p = 0.4880, Chi-squared Test
Statistical Analysis 4: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Percentage of participants with change from baseline at Month 12 in Quality of Life (EQ-5D-Y) being 'Worse'; Test type: Superiority; p = 0.1804, Chi-squared Test

11. Secondary Outcome: Change From Baseline in the Scale for Assessment and Rating of Ataxia (SARA) Score
Description: The SARA included eight items reflecting neurologic manifestations of cerebellar ataxia. The test provides a direct and simple description of motor function in a participant. The test consists of 8 test items: gait, stance, sitting, speech disturbance, finger chase, nose-finger test, fast alternating hand movements, and heel-shin slide. The total score of the 8 items ranges from 0 (normal cerebellar function) to 40 (not able to perform any of the test items).
Time Frame: Baseline to 6 and 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arimoclomol (12-month Double-blind Phase) | Placebo (12-month Double-blind Phase)
Number analyzed (Participants) | 34 | 16
score on a scale
  Change at 6 months | 0.79 [-0.16 to 1.75] | 0.05 [-1.29 to 1.40]
  Change at 12 months | 1.06 [-0.17 to 2.29] | 0.78 [-0.90 to 2.47]
Statistical Analysis 1: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Change from baseline in the SARA score at Month 6 was measured using an ANCOVA model. ANCOVA model was fitted with treatment, baseline SARA score, and use of miglustat as covariates; Test type: Superiority; p = 0.3710, ANCOVA; LS Mean Difference = 0.74, 95% CI 2-sided [-0.92 to 2.40]
Statistical Analysis 2: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Change from baseline in the SARA score at Month 12 was measured using an ANCOVA model. ANCOVA model was fitted with treatment, baseline SARA score and use of miglustat as covariates; Test type: Superiority; p = 0.7899, ANCOVA; LS Mean Difference = 0.28, 95% CI 2-sided [-1.82 to 2.37]

12. Secondary Outcome: Change From Baseline in the Time Spent to Complete the Nine-Hole Peg Test (9HPT)
Description: The 9HPT test is a direct and simple measurement of fine motor coordination function, eye/hand coordination, and the ability to follow a simple direction. The 9HPT is a timed test in which nine pegs are inserted and removed from nine holes in the pegboard. Both hands are tested starting with the dominant hand. The time spent in completing the 9 HPT using each hand was recorded.
Time Frame: Baseline to 6 and 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Arimoclomol (12-month Double-blind Phase) | Placebo (12-month Double-blind Phase)
Number analyzed (Participants) | 34 | 16
seconds
  Dominant Hand: Change at 6 months | 1.54 [-24.98 to 28.06] | 11.88 [-20.88 to 44.64]
  Non-dominant Hand: Change at 6 months | 0.60 [-27.25 to 28.45] | 16.46 [-17.07 to 50.00]
  Dominant Hand: Change at 12 months | -3.29 [-15.56 to 8.98] | -6.49 [-20.34 to 7.37]
  Non-dominant Hand: Change at 12 months | 11.68 [-14.89 to 38.25] | 17.59 [-13.24 to 48.42]
Statistical Analysis 1: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Dominant Hand: Change From Baseline in the Nine-Hole Peg Test (9HPT) at Month 6 was measured using an ANCOVA model: ANCOVA models were fitted with treatment, baseline dominant/non-dominant hand 9HPT time (secs), and use of miglustat as covariates; Test type: Superiority; p = 0.6195, ANCOVA; LS Mean Difference = -10.34, 95% CI 2-sided [-53.01 to 32.33]
Statistical Analysis 2: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Non-dominant Hand: Change From Baseline in the Nine-Hole Peg Test (9HPT) at Month 6 was measured using an ANCOVA model: ANCOVA models were fitted with treatment, baseline dominant/non-dominant hand 9HPT time (secs), and use of miglustat as covariates; Test type: Superiority; p = 0.4693, ANCOVA; LS Mean Difference = -15.87, 95% CI 2-sided [-60.73 to 29.00]
Statistical Analysis 3: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Dominant Hand: Change From Baseline in the Nine-Hole Peg Test (9HPT) at Month 12 was measured using an ANCOVA model: ANCOVA models were fitted with treatment, baseline dominant/non-dominant hand 9HPT time (secs), and use of miglustat as covariates; Test type: Superiority; p = 0.7283, ANCOVA; LS Mean Difference = 3.20, 95% CI 2-sided [-15.71 to 22.12]
Statistical Analysis 4: Comparison: Arimoclomol (12-month Double-blind Phase) vs Placebo (12-month Double-blind Phase); Non-dominant Hand: Change From Baseline in the Nine-Hole Peg Test (9HPT) at Month 12 was measured using an ANCOVA model: ANCOVA models were fitted with treatment, baseline dominant/non-dominant hand 9HPT time (secs), and use of miglustat as covariates; Test type: Superiority; p = 0.7708, ANCOVA; LS Mean Difference = -5.91, 95% CI 2-sided [-47.54 to 35.72]

13. Secondary Outcome: Percentage of Participants Within Each Severity Category of the Clinical Global Impression Scale of Severity (CGI-S)
Description: The CGI-S is a 7-point scale that requires the clinician to rate the severity of the participant's illness at the time of assessment. A rating of 1 is considered normal, or with the least severe symptoms, a rating of 7 is extremely ill, or the worst symptoms. Scores thus range from 1-7 with lower scores indicating less severe disease.
Time Frame: Months 6 and 12
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Arimoclomol (12-month Double-blind Phase) | Placebo (12-month Double-blind Phase)
Number analyzed (Participants) | 29 | 15
percentage of participants
  Month 6: Normal, not ill at all: number analyzed (Participants) | 29 | 14
  Month 6: Normal, not ill at all | 0 | 0
  Month 6: Borderline ill: number analyzed (Participants) | 29 | 14
  Month 6: Borderline ill | 10.3 | 14.3
  Month 6: Mildly ill: number analyzed (Participants) | 29 | 14
  Month 6: Mildly ill | 27.6 | 28.6
  Month 6: Moderately ill: number analyzed (Participants) | 29 | 14
  Month 6: Moderately ill | 10.3 | 35.7
  Month 6: Markedly ill: number analyzed (Participants) | 29 | 14
  Month 6: Markedly ill | 31.0 | 0
  Month 6: Severely ill: number analyzed (Participants) | 29 | 14
  Month 6: Severely ill | 20.7 | 14.3
  Month 6: Most extremely ill participants: number analyzed (Participants) | 29 | 14
  Month 6: Most extremely ill participants | 0 | 7.1
  Month 12: Normal, not ill at all: number analyzed (Participants) | 27 | 15
  Month 12: Normal, not ill at all | 0 | 0
  Month 12: Borderline ill: number analyzed (Participants) | 27 | 15
  Month 12: Borderline ill | 7.4 | 6.7
  Month 12: Mildly ill: number analyzed (Participants) | 27 | 15
  Month 12: Mildly ill | 29.6 | 26.7
  Month 12: Moderately ill: number analyzed (Participants) | 27 | 15
  Month 12: Moderately ill | 11.1 | 33.3
  Month 12: Markedly ill: number analyzed (Participants) | 27 | 15
  Month 12: Markedly ill | 29.6 | 6.7
  Month 12: Severely ill: number analyzed (Participants) | 27 | 15
  Month 12: Severely ill | 22.2 | 26.7
  Month 12: Most extremely ill participants: number analyzed (Participants) | 27 | 15
  Month 12: Most extremely ill participants | 0 | 0

14. Secondary Outcome: Percentage of Participants Within Each Category of the Clinical Global Impression Scale of Improvement (CGI-I)
Description: The CGI-I is a 7-point scale that rates total improvement of participant's condition. The clinician rates the participants from 1=Very much improved, 2=Much improved, 3=Minimally improved, 4=No change, 5=Minimally worse, 6=Much worse, or 7=Very much worse. Scores thus range from 1-7 with lower scores indicating greater improvement.
Time Frame: Months 6 and 12
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Arimoclomol (12-month Double-blind Phase) | Placebo (12-month Double-blind Phase)
Number analyzed (Participants) | 29 | 15
percentage of participants
  Month 6: Very Much Improved: number analyzed (Participants) | 29 | 12
  Month 6: Very Much Improved | 3.4 | 0
  Month 6: Much Improved: number analyzed (Participants) | 29 | 12
  Month 6: Much Improved | 0 | 0
  Month 6: Minimally Improved: number analyzed (Participants) | 29 | 12
  Month 6: Minimally Improved | 24.1 | 25.0
  Month 6: No Change: number analyzed (Participants) | 29 | 12
  Month 6: No Change | 37.9 | 25.0
  Month 6: Minimally Worse: number analyzed (Participants) | 29 | 12
  Month 6: Minimally Worse | 27.6 | 33.3
  Month 6: Much Worse: number analyzed (Participants) | 29 | 12
  Month 6: Much Worse | 6.9 | 16.7
  Month 6: Very Much Worse: number analyzed (Participants) | 29 | 12
  Month 6: Very Much Worse | 0 | 0
  Month 12: Very Much Improved: number analyzed (Participants) | 27 | 15
  Month 12: Very Much Improved | 0 | 0
  Month 12: Much Improved: number analyzed (Participants) | 27 | 15
  Month 12: Much Improved | 3.7 | 6.7
  Month 12: Minimally Improved: number analyzed (Participants) | 27 | 15
  Month 12: Minimally Improved | 18.5 | 33.3
  Month 12: No Change: number analyzed (Participants) | 27 | 15
  Month 12: No Change | 51.9 | 20.0
  Month 12: Minimally Worse: number analyzed (Participants) | 27 | 15
  Month 12: Minimally Worse | 14.8 | 13.3
  Month 12: Much Worse: number analyzed (Participants) | 27 | 15
  Month 12: Much Worse | 7.4 | 26.7
  Month 12: Very Much Worse: number analyzed (Participants) | 27 | 15
  Month 12: Very Much Worse | 3.7 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to last dose of blinded study treatment (Month 12)
Description: Safety analysis set included all participants who had received at least one dose of study drug. Adverse events were reported separately for the single dose period where 28 participants less than 12 years old received a single dose of arimoclomol, and the 12-month continuous dose period where all participants received randomized treatment.
Arm/Group | Arimoclomol Single PK Dose | Arimoclomol (12-month Double-blind Phase) | Placebo (12-month Double-blind Phase)
All-Cause Mortality (participants affected / at risk) | 0/28 | 1/34 | 0/16
Serious Adverse Events (participants affected / at risk) | 2/28 | 5/34 | 6/16
Other Adverse Events (participants affected / at risk) | 4/28 | 30/34 | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arimoclomol Single PK Dose (N=28) | Arimoclomol (12-month Double-blind Phase) (N=34) | Placebo (12-month Double-blind Phase) (N=16)
Cardio-respiratory Arrest (Cardiac disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 2
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 2
Epileptic Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Aspiration Bronchial (Investigations) | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arimoclomol Single PK Dose (N=28) | Arimoclomol (12-month Double-blind Phase) (N=34) | Placebo (12-month Double-blind Phase) (N=16)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 6 | 3
Drug Hypersensitivity (Immune system disorders) | 1 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 6 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1 | 0
Deafness Neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0
Deafness Unilateral (Ear and labyrinth disorders) | 0 | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Pupils Unequal (Eye disorders) | 0 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0
Aphthous Ulcer (Gastrointestinal disorders) | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 7 | 3
Dental Caries (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 7 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 1
Lip Dry (Gastrointestinal disorders) | 0 | 1 | 0
Mouth Cyst (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0
Salivary Hypersecretion (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 8 | 4
Asthenia (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 0
Gait Disturbance (General disorders) | 0 | 1 | 0
Medical Device Site Dermatitis (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0
Peripheral Swelling (General disorders) | 0 | 1 | 0
Secretion Discharge (General disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic Lesion (Hepatobiliary disorders) | 0 | 1 | 0
Food Allergy (Immune system disorders) | 0 | 1 | 0
Seasonal Allergy (Immune system disorders) | 0 | 2 | 1
Bronchitis (Infections and infestations) | 0 | 4 | 2
Conjunctivitis (Infections and infestations) | 0 | 1 | 1
Ear Infection (Infections and infestations) | 0 | 0 | 2
Eye Infection (Infections and infestations) | 0 | 0 | 2
Fungal Infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 2
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1
Hand-foot-and-mouth Disease (Infections and infestations) | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 1
Localised Infection (Infections and infestations) | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 3 | 0
Medical Device Site Infection (Infections and infestations) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 4
Onychomycosis (Infections and infestations) | 0 | 1 | 0
Oral Candidiasis (Infections and infestations) | 0 | 1 | 0
Oral Fungal Infection (Infections and infestations) | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 3 | 1
Rhinitis (Infections and infestations) | 0 | 5 | 2
Skin Candida (Infections and infestations) | 0 | 1 | 0
Viral Infection (Infections and infestations) | 0 | 1 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Eschar (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tooth Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood Creatinine Increased (Investigations) | 0 | 1 | 0
Body Temperature Abnormal (Investigations) | 0 | 0 | 1
Body Temperature Increased (Investigations) | 0 | 1 | 0
C-reactive Protein Increased (Investigations) | 0 | 1 | 0
Vitamin D Decreased (Investigations) | 0 | 1 | 0
Weight Decreased (Investigations) | 0 | 5 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 3 | 0
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Refeeding Syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Vitamin C Deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 3 | 1
Lethargy (Nervous system disorders) | 0 | 2 | 0
Memory Impairment (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Motor Dysfunction (Nervous system disorders) | 0 | 1 | 0
Muscle Spasticity (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Peroneal Nerve Palsy (Nervous system disorders) | 0 | 1 | 0
Petit Mal Epilepsy (Nervous system disorders) | 0 | 1 | 0
Quadriplegia (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 3 | 1
Speech Disorder (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 2 | 0
Aggression (Psychiatric disorders) | 0 | 2 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 1 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 1 | 0
Sleep Disorder (Psychiatric disorders) | 0 | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 1 | 0
Premenstrual Syndrome (Reproductive system and breast disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dandruff (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Henoch-Schonlein Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Gastrostomy (Surgical and medical procedures) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Cataplexy (Nervous system disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT02612129/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT02612129/SAP_001.pdf